CLINICAL TRIAL: NCT03218254
Title: MethylphenIdate for Fatigue in Haematological Cancer. A Randomized, Double-blind, Placebo-controlled, CROssover Trial - the MICRO Trial
Brief Title: MethylphenIdate for Fatigue in Haematological Cancer
Acronym: MICRO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henrik Frederiksen (Other)
Responsible Party: Sponsor-Investigator, Henrik Frederiksen, Professor, MD, PHD, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EUDRACT 2017-001844-36
Record Dates: First submitted 2017-07-13; First posted 2017-07-14 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Hematological Cancer
Keywords: hematological cancer, fatigue, quality of life
MeSH Terms: conditions — Fatigue | interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: Methylphenidate or Placebo titrated according to effect and toxicity week 1-6 followed by 1 week of washout and then crossover followed by repeated procedures with the other treatment for week 8-13.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical placebo tablets are produced. Study pharmacy produces study medication containers and randomizes patients, and keeps track of unique study IDs. Unblinding is only done after completion or in emergency situations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylphenidate - Placebo (Other): Methylphenidate before placebo
  Interventions: Drug: Methylphenidate; Drug: Placebo
- Placebo - Methylphenidate (Other): Methylphenidate after placebo
  Interventions: Drug: Methylphenidate; Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — Titration of MTP for treatment of fatigue
Drug: Placebo — Placebo

SUMMARY:
Cancer related fatigue (CRF) is the most debilitating problem for patients with haematological cancer. CRF severely reduces quality of life (QoL), functional capacity, impacts health behavior, recovery and furthermore no approved treatment exists. In solid cancer methylphenidat (MTP) has been suggested to improve CRF, however patients with haematological cancer has not been studied. The current randomized placebo controlled study includes a variety of severely fatigued haematological cancer patients from seven Danish departments. It aims at revealing whether MTP can improve CRF, functional capacity and QoL thereby hopefully providing improvement and treatment options in this field where improvements are requested the most by patients. Patients are randomized to treatment with MTP or placebo week 1-6 followed by "wash-out" and cross-over - placebo to MTP or vice versa - during week 8-13. End-points will be patient reported fatigue, as well as improvements in active hours, functional capacity, and QoL.

DETAILED DESCRIPTION:
BACKGROUND Survival prognosis in haematological malignancies has improved considerably, however the frequency and impact of the most prevalent and debilitating symptoms - cancer related fatigue (CRF) - has not improved. Up to 40% of cancer patients has daily difficulties due to CRF and fatigue and weakness is affecting 2/3 of patients. In contrast to everyday fatigue CRF is defined as an unusual and persistent sense of tiredness, weakness, or even exhaustion that is not relieved by rest or sleep and leads to decreased physical or mental capacity.

Haematological cancer is often associated with fatigue due to both anemia and constitutional symptoms. Myeloablative chemotherapeutic regimens and stem cell transplantations are unique for haematological cancer treatment and these very potent regimens may result in CRF even after several years. CRF among haematological cancer patients is associated with reduced adherence to physicians recommendations [11] and permanent withdrawal from labor market. Patients express that their single most prevalent and severe problem is "dealing with feeling tired", exceeding the proportion who expresses problems "in dealing with not feeling sure that the cancer has gone" or "being told they had cancer".

An increasing emphasis has been given to rehabilitation in cancer patients and individualized exercise programs; however, these will only be feasible among a minority of haematological cancer patients. In recent years, studies using methylphenidate (MTP) in the treatment of CRF in solid cancer have been conducted, some of which have found improvements in fatigue with MTP and without significant adverse effects. These studies show that MTP may be beneficial in management of CRF. However, patients in concurrent chemotherapy were unlikely to benefit.

STUDY RATIONALE AND OBJECTIVE Patients with haematological malignancies have a severe unmet need in dealing with CRF and hardly any patients with haematological malignancies have been included in previous intervention studies. MTP treatment has been found to be safe in this setting . The current study aims at studying whether MTP can be used for management of CRF in patients with haematological cancer in order to improve also functional capacity and quality of life (QoL). Many of the patients in the current study will have no other treatment options to improve their fatigue, QoL, and functional capacity.

STUDY END-POINTS The primary end point it patient reported fatigue after six weeks of MTP treatment measured by the FACIT-F scale. A good clinical response is defined as a 25% reduction in fatigue from baseline score. Secondary end-points are changes in hours awake, in time spend at work, being social, house work / gardening, being outside, participating in exercise, in muscle strength and endurance, in QoL, and in number of blood transfusions.

STUDY POPULATION AND DESIGN The study population comprises 150 patients with haematological malignancies who are not in current chemotherapy. The patients will be included from seven haematological out-patient clinics in Denmark. The haematological out-patient clinics have a large group of chronic severely fatigued haematological cancer patients that will be approached for inclusion in the trial. Power calculations, and assumptions behind as well as a detailed list of inclusion and exclusion criteria are available from full study protocol.

Patients will be randomized (1:1) to MTP or placebo treatment for 6 weeks. After this time points patients treated with MTP will after one week wash-out cross over to placebo treatment and vice versa (Figure). The rationale for the crossover design is that the study includes a variety of different haematological malignancies with different symptomatology, course, management and different degree of bone-marrow failure. When using patients as their own controls the effects of these factors are accounted for. Treatment will be blinded to the patient, treating investigators, staff, sponsor, and study secretariat. Patients will be randomized to start either MTP or matching placebo twice daily. The dosage will start at 5 mg twice daily at 8 am and 1 pm or matching placebo and can be titrated to a maximum of 20mg twice daily or matching placebo. From day 1 in week 8 treatments will be crossed over from either MTP to placebo or vice versa (Figure).

FATIGUE AND QUALITY OF LIFE ASSESSMENT TOOLS The fatigue assessment scale - FACIT-F - has been widely used in studies of cancer related fatigue and a FACIT-F score change both as a covariate and as the main outcome measure in interventional studies. In line with us previous clinical trials used a single VAS-fatigue assessment for inclusion prior to treatment. The visual analogous scale is 100 mm long and ranges from 0 = "not tired" to 10 = "worst possible tiredness". The European Organisation for Research and Treatment of Cancer (EORTC) QoL questionnaires are among the most widely used tools for assessing physical and psychosocial symptoms in cancer patients. The EORTC-QLQ-C15-PAL was developed for the palliative setting [24]. Permission to include the fatigue and QoL scales has been granted to the trial.

EFFICACY EVALUATION Efficacy of MTP treatment will be evaluated using FACIT-F, EORTC-QLQ-C15-Pal, VAS-F as well as patients' perception on their energy and diaries on activities. The study is powered to show a 4.25 point reduction in the FACIT-F scale (corresponding to an estimated 25% reduction from baseline) that has been suggested as a minimal important difference in studies of CRF. Assessments of functional capacity (muscle strength and endurance) as well as patients' actual daily chores are also included in this evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Malignant haematological disease such as

  * Myeloproliferative neoplasm
  * Myelodysplasia / Acute Myeloid Leukemia / Chronic Myelomonocytic leukemia
  * Acute lymphoblastic leukemia
  * Malignant lymphoma
  * Chronic lymphocytic leukemia
  * Multiple myeloma
* Patient reported fatigue equals to a VAS score of 4 or more on a scale of 0 to 10 on (0 = no fatigue to 10 = worst possible fatigue). Score must be the patients retrospective estimate of usual fatigue during the past two weeks
* Out-patient at inclusion
* Hb ≥ 5 mmol/l on the past three hb measurements
* Age ≥ 18 years
* Ability to read and understand Danish language
* Safe contraception for fertile women

Exclusion Criteria:

* Chemotherapy within last 8 weeks. Patients on a stable dose previous 4 weeks of the following, may be included:

  * Kinase inhibitors (such as Imatinib, Dasatininb, Nilotinib, Ruxulitinib, Bosutinib and others)
  * Hydroxyurea
  * Chlorambucil
  * Busulfan
  * Melphalan
  * alfa-interferon
  * IMIDs (such Thalidomide, Lenalidomide, Pomalidomide and others)
  * monoclonal anti-bodies
  * 5-azacytidin
  * Combinations of above mentioned drugs and with corticosteroids (CS) are allowed as long as CS dose restrictions are followed.
* Glucocorticoid treatment exceeding the equal of prednisolone 10mg / day or equivalent average dose / week and dosage must have remained stable during the past 4 weeks.
* Current infection
* Previous or current diagnosis made by a psychiatrist of psychosis, mania, or Tourette
* Known previous suicidal attempts
* Current psycho-pharmacological treatment
* Known cardio-vascular disease. Patients with known stable angina pectoris may be included.
* Prolonged QT interval corrected (QTc) >500msec at screening ECG
* Known cerebro-vascular disease
* Uncontrolled hypertension defined as SBP > 160 mmHg or DBP > 100mmHg
* Cognitive impairment as judged by investigator
* Change in opiod dose during the past two weeks
* Life expectancy < 4 months
* EPO started or dosage changed < 6 weeks prior to inclusion
* Hypothyroidism with thyroid hormone supplementation treatment started or dosage changed < 6 weeks before inclusion
* Known hyperthyroidism
* Known pheochromocytoma
* Known glaucoma
* Previous or current substance abuse
* Use of monoamine oxidase inhibitors within last two weeks
* Known allergy to or side-effects from previous methylphenidate treatment
* Pregnancy or breast feeding
* Serious medical illness which in the judgement of the investigator would make the patient inappropriate for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-06-08 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue score | end of 6th or 13th week

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided